CLINICAL TRIAL: NCT02745418
Title: Deconstructing the Atopic March - the Role of Filaggrin Mutations and Sensitization Pathways in Allergic Rhinitis and Peanut Allergy
Brief Title: The Role of Filaggrin Mutations and Sensitization Pathways in Allergic Rhinitis and Peanut Allergy
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Anne Ellis (Other)
Responsible Party: Sponsor-Investigator, Dr. Anne Ellis, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: FLG-AR-001
Record Dates: First submitted 2016-03-02; First posted 2016-04-20 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Allergic Rhinitis; Peanut Allergies
MeSH Terms: conditions — Rhinitis, Allergic; Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected and DNA will be isolated for genotyping of filaggrin mutations.
Oversight: Data Monitoring Committee: No

SUMMARY:
Caucasian male and female participants age 18 years of age and older will be enrolled in this study if they have known birch or peanut allergies or known to be non-atopic. Participants will undergo skin testing to confirm their allergies if not completed in the last 12 months. Medications and medical history will be captured with a focus on atopic disorders. Participants will undergo birch and peanut patch testing to assess penetration and if potential correlation exists with filaggrin genotyping and phenotyping. Blood samples will be drawn from participants and DNA isolated for genotyping of null mutations in filaggrin.

DETAILED DESCRIPTION:
Participants with confirmed history of birch induced allergic rhinitis or peanut allergy or that are non-atopic will undergo the following procedures.

If not already completed in the previous year, participants will be skin tested to a panel of common environmental allergens, including birch pollen and peanut. To be considered "non-atopic", all skin tests in the panel must be negative in the presence of a positive histamine control. All participants will also be skin tested to peanut, Arah 2, Ara h 8 (if obtainable), crushed raw unroasted peanut, peanut butter, peanut extract, Bet v 1 and birch pollen extract.

Blood samples will be drawn for genotyping of the four most common null mutations in FLG in Caucasians (R501X, 2282del4, R2447X, S3247X).

Patch testing will be performed using Ara h2, Arah8 (if obtainable), crushed raw unroasted peanut, peanut butter, peanut extract, Bet v 1 and birch pollen extract. Peanut and birch pollen allergens, both whole and components will be diluted 1:10 in both saline and petroleum jelly and applied to normal controls skin to establish levels for irritant reaction. If further dilutions are required to show non-irritation these will be performed.

As well, a limited medical history and medication history will be documented, with a focus on atopic disorders (i.e. atopic dermatitis (eczema), allergic rhinitis, asthma, and food allergy). Those in the non-allergic control group will be excluded if they have features of eczema, food allergy or other atopic conditions). Medications that could potentially interfere with the skin test results (i.e. antihistamines) must be documented, and appropriate washout intervals observed prior to the skin test procedure, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* caucasian male or females
* participants 18 years of age and older
* participants with known birch allergy, confirmed by a skin test 3mm or greater than the negative control
* participants with diagnosed and confirmed peanut with allergy
* confirmed by one of the following:
* positive food challenge
* convincing history of peanut allergy AND positive skin test (3mm >= than negative control) OR peanut-specific IgE >=0.35
* uncertain history of peanut allergy OR no exposure to peanut AND a positive skin test 5mm>= negative control AND a peanut-specific IgE >=15
* non-allergic controls who lack a diagnosis of any atopic diathesis and have supportive negative skin testing to a panel of common environmental allergens.

Exclusion criteria:

* participants unable to complete study related procedures
* participants that have taken or are taking restricted medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian male and female participants 18 years of age and older with birch or peanut allergies as well as non-atopic controls will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Peanut patch testing | Up to 17 months
  Differences in patch test positive responses to peanut allergen (extract plus raw peanut butter preparations) between participants with confirmed peanut allergy, confirmed birch allergy and non-atopic controls.
  Responses are graded as:
  Negative (-) Irritant reaction (IR) Equivocal / uncertain (+/-) Weak positive (+) Strong positive (++) Very Strong Positive (+++)

SECONDARY OUTCOMES:
Birch patch testing | Up to 17 months
  Differences in patch test positive responses to birch allergen extract between participants with confirmed peanut allergy, confirmed birch allergy and non-atopic controls.
  Responses are graded as:
  Negative (-) Irritant reaction (IR) Equivocal / uncertain (+/-) Weak positive (+) Strong positive (++) Very Strong Positive (+++)

OTHER OUTCOMES:
Relationship of peanut and birch patch testing responses to filaggrin genotype | Up to 17 months
  Presence or absence of positive patch tests to birch and peanut and correlation of these responses with filaggrin genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No